CLINICAL TRIAL: NCT06069635
Title: Effect of Fatigue on Core Endurance, Dynamic Balance and Player Performance in Adolescent Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Rageh Saber Ali, Assistant lecturer, Badr University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RageH1
Record Dates: First submitted 2023-09-27; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Fatigue
Keywords: core endurance; football; balance
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fatigue group (Experimental): 30 male players will be assessed for core endurance, balance and performance then fatigue protocol will be applied and measure for core endurance, balance and performance after fatigue
  Interventions: Other: Fatigue protocol (repeated sprint ability)
- Control group (Sham Comparator): 30 players will be assessed for core endurance, balance and performance. Players will be assessed at baseline then take rest drink water and then measure for core endurance, balance and performance again .
  Interventions: Other: Sham Comparator: Control group

INTERVENTIONS:
Other: Fatigue protocol (repeated sprint ability) — The test performed on an outdoor field (artificial grass carpet) in the form of 6 repetitions of maximal 2× 15 m shuttle sprints interspersed with 20 seconds of passive recovery , Before the RSA protocol, all players perform a brief standardized warm-up (approximately 20 minutes long), in 1at submaximal speed (followed by 40 seconds of passive recovery The fatigue index (FI) used to characterize the RSA performance was calculated in terms of percentage decrement score At the end of the RSA protocol , usually the time elapsed between the end of the last sprint and the beginning of the measurements was no more than 20 seconds, to avoid masking effects related to progressive recovery from fatigue.
  Arms: Fatigue group
Other: Sham Comparator: Control group — approximately 20 minutes long), which consisted of : 6 minutes of incremental running from 60% to 80% of maximal aerobic speed; 6 minutes of dynamic flexibility exercises; 2 minutes of forward, backward, and lateral jogging and high-knee and ''butt-kick'' runs; 2 minutes of shuttle sprints (5 m in 1 direction and 5 m in the opposite direction, repeated for 2 minutes) at submaximal speed (followed by 40 seconds of passive recovery); and 2 minutes of RSA protocol simulation at submaximal speed (2 repetitions), again followed by 40 seconds of passive recovery. take apenalty of water and rest
  Arms: Control group

SUMMARY:
The goal of this clinical study is to investigate the effect of fatigue on balance, core endurance and player performance in adolescent football players. the main questions it aims to answer are:

1. What is the effect of fatigue on balance, core endurance and player performance in adolescent football players?
2. What is the effect of balance on player performance in adolescent football players? participants will be 60 male age from 16 to 18 years selected from Wadi-Degla football club randomly assigned into either fatigue or control group, Each player assessed for core endurance, balance and performance then fatigue protocol applied for the fatigue group and shame protocol for the control group and the repeat all measurements.

DETAILED DESCRIPTION:
This study will be conducted in This pre and post controlled trial aiming at determining the efficacy of fatigue on core endurance, balance and player performance in adolescent football players, this study will be conducted in Wadi-Degla football club.

Players will be randomly assigned into either fatigue or control group. Randomizations will be done using computer random generated numbers.

Fatigue group (F.G): 30 players will be assessed for core endurance, balance and performance then fatigue protocol will be applied and reasses for core endurance, balance and performance after fatigue Control Group (C.G): 30 players will be assessed for core endurance, balance and performance.

Players will be assessed at baseline and fatigue for: balance using (MFT challenge disc),Core endurance, 20-m running sprint and Triple-Hop Test (THT) for perfprmace Will apply RSA as fatigue protocol for the fatigue groupe.

Inclusion criteria:

Players will be included according to the eligibility Criteria

ELIGIBILITY:
Inclusion Criteria:

1. age ranges from 14 to 18 years old
2. Players will selected from Wadi-Degla (2005, 2006 and 2007 football teams )
3. All participants will be free from lower limb injuries for at least 6 months before the study
4. Body mass index will be at optimal (18.5 to 24.9)

Exclusion Criteria:

1. Not regularly trained for at least 6 hours per week
2. Major lower limb injuries for at least 6 months before the study.
3. lower limb surgery for before the study

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2023-06-17 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
single-leg balance test | 20 seconds
  The "MFT challenge disc" balance measuring system will be used to assess single-leg balance test (SLBT) for both the dominant (D) and non-dominant (N) legs (i.e., SLBT-D, SLBT-N).

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed sh Abdelsalam, phd, Study Chair — Cairo University; Mona se Mohamed, phd, Study Director — Badr University; Karim mo Fawzy, phd, Study Director — Cairo University
Locations (1):
- Cairo University, Giza, Egypt